CLINICAL TRIAL: NCT01322295
Title: Human Bronchial Microdialysis in Open Aortic Aneurysm Repair
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/1649a
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elective open aortic aneurysm repair has an overall reported 30 day mortality of 2-6 percent, but in patients more than 65-70 years the mortality is reported to be more than 10 percent. The phenomenon of acute lung injury (ALI)/adult respiratory distress syndrome (ARDS) after infra renal abdominal aneurysm repair caused by ischemia-reperfusion is well established. The degree of disability varies from a light degree of acute respiratory failure to mortality for patients with the same profile of risk.

Primary aim is to develop a model that monitors inflammatory marker molecules collected from the bronchial epithelial lining fluid by microdialysis. The method with examination of the bronchial epithelial lining fluid by microdialysis and analysis of multiple inflammation markers as previously done by the investigators group.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned for elective open aortic surgery

Exclusion Criteria:

* Moderate to severe COPD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients assigned for elective open aortic surgery are enrolled by invitation
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cytokines in bronchial epithelial lining fluid | Within 4 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erik Solligård, md phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Tyvold SS, Solligard E, Gunnes S, Lyng O, Johannisson A, Gronbech JE, Aadahl P. Bronchial microdialysis of cytokines in the epithelial lining fluid in experimental intestinal ischemia and reperfusion before onset of manifest lung injury. Shock. 2010 Nov;34(5):517-24. doi: 10.1097/SHK.0b013e3181dfc430. PMID 20354465
- [Result] Tyvold SS, Dahl T, Dragsund S, Gunnes S, Lyng O, Damas JK, Aadahl P, Solligard E. Bronchial microdialysis monitoring of inflammatory response in open abdominal aortic aneurysm repair; an observational study. Physiol Rep. 2017 Jul;5(14):e13348. doi: 10.14814/phy2.13348. PMID 28743822